CLINICAL TRIAL: NCT02305108
Title: Evaluation of the Efficacy of Treatment of the Soft Tissues With Fascial Manipulation for Patients That Are Waiting for Total Hip Arthroplasty in Osteoarthritis
Brief Title: Fascial Manipulation in Patients With Hip Osteoarthritis
Acronym: manifahip
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Prot. gen. 0018810
Record Dates: First submitted 2014-09-30; First posted 2014-12-02 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-08

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- fascial manipolation and standard (Experimental)
  Interventions: Other: fascial manipulation; Other: standard treatment
- standard treatment (Active Comparator)
  Interventions: Other: standard treatment

INTERVENTIONS:
Other: fascial manipulation — Recruited patients in study's group will be treated with the standard treatment and fascial manipulation.
  Specific points of fascial tissue will be treated with a deep friction to improve elasticity.
  The number of point treated will be refered to a specific evaluation for each patient.
  Fascial manipulation provide 3 session treatment (one treatment for week).
  Arms: fascial manipolation and standard
Other: standard treatment — Before surgery, standard physiotherapy treatment provides an education session about the rehabilitation program tha is going to be execute after surgery.
  After surgery 2 daily physiotherapy treatment are implemented: bed exercise as active and passive flex-extension of lower limb, movements for postural change to reach sitting and standing position, walking training.

SUMMARY:
The study will test the efficacy of the treatment of soft tissues for osteoarthritis patients that are waiting for total hip arthroplasty. The fascial manipulation provides a deep pressure of specific points of the muscle fascia. The aims of this treatment are the improve of pain before the surgery and the improve of functional performance after the surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients age 40-80, with primary coxarthrosis waiting for total hip arthroplasty that complain a pain measured by Numeric Rating Scale ≥ 5 and that live in Bologna

Exclusion Criteria:

* arthroplasty revision or substitution. Patient with cognitive deficiency and severe comorbidity (rheumatic, neurological or cardiovascular pathology)

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-06; Primary Completion 2015-05 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
pain is measured by numeric rating scale | 3 weeks before surgery

SECONDARY OUTCOMES:
performance measurement assessed with Oxford Hip Scale, 30 second chair stand test, 10 meters walking test, Iova level of assistance. | a month after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Cotti, PT, Principal Investigator — Istituto Ortopedico Rizzoli
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Bo, Italy